CLINICAL TRIAL: NCT04573673
Title: Efficacy and Safety of Transcutaneous Tibial Neuro-stimulation to Improve Voiding Dysfunction in Multiple Sclerosis Patients.
Brief Title: Transcutaneous Tibial Neuro-stimulation to Improve Voiding Dysfunction in Multiple Sclerosis.
Acronym: NEUROSTIM-SEP1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018_27; 2018-A03045-50 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis; Lower Urinary Tract Symptoms
Keywords: Multiple sclerosis; Voiding dysfunction; Bladder-sphincter dyssinergia; Tibial neuro-stimulation
MeSH Terms: conditions — Multiple Sclerosis; Lower Urinary Tract Symptoms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTNS verum (Experimental): Patients will be treated with transcutaneous tibial neuro-stimulation with one 30-minute session daily for a period of 12 weeks.
  Interventions: Device: PTNS de verum
- PTNS placebo (Sham Comparator): Patients will be treated with placebo (i.e. no current) transcutaneous tibial neuro-stimulation for 30 consecutive minutes daily for 12 weeks (same treatment regimen as the experimental group).
  Interventions: Device: PTNS placebo

INTERVENTIONS:
Device: PTNS de verum — The device will be set to program P-4: Frequency 20Htz, Pulse duration = 200 µs. The amplitude (Volt) will be adjusted by the patient according to the feeling.
  Other Names: Peristim Pro (CEFAR-COMPEX®)
  Arms: PTNS verum
Device: PTNS placebo — The device will be set to program P-4: Frequency 20Htz, Pulse duration = 200 µs. A resistor will be incorporated in the device to block the passage of electric current
  Other Names: Peristim Pro (CEFAR-COMPEX®
  Arms: PTNS placebo

SUMMARY:
The present trial is designed to assess the efficacy and safety of transcutaneous tibial neuro-stimulation (TTNS) in improving bladder emptying in multiple sclerosis (MS) patients.

Patients presenting with MS and performing clean intermittent self-catheterization (CISC) to empty the bladder in the context of voiding dysfunction, will be eligible.

Included patients will be randomly assigned to two distinct arms

* PTNS de verum : patients will be treated with transcutaneous tibial neuro-stimulation at a rate of one session of 30 consecutive minutes daily for a period of 12 weeks.
* PTNS placebo : Patients will be treated with placebo (i.e. no current) transcutaneous tibial neuro-stimulation for 30 consecutive minutes daily for a period of 12 weeks (same treatment regimen as the experimental group).

Efficacy in improving voiding dysfunction will be assessed 12 weeks after randomization using the BVE ratio (Bladder Voiding Efficiency) = Ratio of urine volume / total bladder volume.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of multiple sclerosis
* Patient with bladder-sphincter dyssinergia
* Patient using clean intermittent self-catheterization as exclusive bladder management
* Patient who has given written consent
* Socially insured patient
* Patient willing to comply with all study procedures and study duration

Exclusion Criteria:

* Patient with other associated neurological pathology
* Patient with an Expanded Disability Status Scale (EDSS) score ≥ 6
* Patient with recurrent urinary tract infections (> 3 episodes / year)
* Patient with uncontrolled overactive bladder
* Patient with uncontrolled detrusor hyperactivity
* Patient with a bladder compliance disorder
* Patient with tibial neuro-stimulation in the last 3 months
* Patient treated with a sacral neuro-modulation
* Patient who has received an intradermal injection of botulinum toxin A within the last 9 -months Patient who received alpha-blocker treatment within the last month Patient with benign prostatic hypertrophy (prostate volume > 40 cc) - Last ultrasound scan < 6 months.

Patient with one or more bladder diverticulum(s) Patient with unilateral or bilateral renal Patient with unilateral or bilateral vesico-ureteral reflux Patient with impaired renal function (GFR according to CKD-EPI < 60 ml/min/1.73m2) Patient with a metallic prosthesis on the lower limb Patient with a Pacemaker Pregnant patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
BVE ratio (Bladder Voiding Efficiency) = Ratio of urine volume / total bladder volume | At 12 weeks after randomization
  BVE will be measured during the multi-channel urodynamic study

SECONDARY OUTCOMES:
Maximal flow rate (mL/s) on multi-channel urodynamic study | At baseline, At 12 weeks after randomization
  Maximal flow rate will be measured during the multi-channel urodynamic study
Post-void residual volume (mL) on multi-channel urodynamic study | At 12 weeks after randomization
  Post-void residual volume will be measured during the multi-channel urodynamic study
Maximal detrusor pressure during micturition (cmH2O) on multi-channel urodynamic study | At 12 weeks after randomization
  Maximal detrusor pressure during micturition will be measured during the multi-channel urodynamic study
Mean voided volume (mL) on a three-day ambulatory measure | At 12 weeks after randomization
  Mean voided volume will be measured using an ambulatory flowmeter (Homeflow®) during three consecutive days
Mean maximal flow rate (mL/s) on a three-day ambulatory measure | At 12 weeks after randomization
  Mean maximal flow rate will be measured using an ambulatory flowmeter (Homeflow®) during three consecutive days
Mean post-void residual volume (mL) on a three-day ambulatory measure | At 12 weeks after randomization
  Mean post-void residual volume will be measured using an ambulatory flowmeter (Homeflow®) during three consecutive days.
Frequency of patients who were able to stop clean intermittent self-catheterization (PVR < 100 mL) | At 12 weeks after randomization
  Mean post-void residual volume will be measured using an ambulatory flowmeter (Homeflow®) during three consecutive days
Urinary symptoms self-reported questionnaire (USP) | At 12 weeks after randomization
  USP : Urinary Symptom Profile
Quality of life self-reported questionnaire (Qualiveen) | At 12 weeks after randomization
  Qualiveen
Difficulty to perform CISC self-reported questionnaire (ICDQ) | At 12 weeks after randomization
  ICDQ : Intermittent Catheterization Difficulty Questionnaire
Digestive symptoms self-reported questionnaire (NBD) | At 12 weeks after randomization
  NBD : Neurogenic Bowel Dysfunction
Digestive symptoms self-reported questionnaire (Wexner) | At 12 weeks after randomization
  Wexner questionnaire
Sexual symptoms self-reported questionnaire (FSFI) | At 12 weeks after randomization
  FSFI (female) : Female Sexual Function Index
Sexual symptoms self-reported questionnaire ( MSHQ) | At 12 weeks after randomization
  MSHQ (male) : Male Sexual Health Questionnaire
Frequency of patients with detrusor overactivity on multi-channel urodynamic study | At 12 weeks after randomization
  Detrusor overactivity will be objectify during the multi-channel urodynamic study
Filling volume (mL) at first detrusor unhibited contraction on multi-channel urodynamic study - If detrusor overactivity. | At 12 weeks after randomization
  Filling volume at first detrusor unhibited contraction will be measured during the multi-channel urodynamic study.
Maximal detrusor pressure (cmH2O) on multi-channel urodynamic study - If detrusor overactivity. | At 12 weeks after randomization
  Maximal detrusor pressure will be measured during the multi-channel urodynamic study
Maximal cystomanometric capacity (cmH2O) on multi-channel urodynamic study | At 12 weeks after randomization
  Maximal cystomanometric capacity will be measured during the multi-channel urodynamic study
Frequency of adverse events occurring during the 12-week follow-up | Measured 12 weeks after randomization
  Adverse events will be exhaustively listed

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Biardeau, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France